CLINICAL TRIAL: NCT05204563
Title: A Multicenter, Randomized, Double-Blind, Comparative, Phase 3 Study to Evaluate the Efficacy and Safety of Intravenous Imipenem/Cilastatin/XNW4107 in Comparison With Imipenem/Cilastatin/Relebactam in Adults With Hospital-Acquired Bacterial Pneumonia or Ventilator-Associated Bacterial Pneumonia (EudraCT no. 2022-000081-18) (EUCTR no. 2022-501952-27-00) (IND no. 146614)
Brief Title: Imipenem/Cilastatin-XNW4107 Versus Imipenem/Cilastatin/Relebactam for Treatment of Participants With Bacterial Pneumonia (XNW4107-302, REITAB-2)
Acronym: REITAB-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Evopoint Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XNW4107-302
Record Dates: First submitted 2022-01-05; First posted 2022-01-24 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Hospital Acquired Bacterial Pneumonia or Ventilator-Associated Bacterial Pneumonia
MeSH Terms: interventions — Cilastatin; imipenem, cilastatin and relebactam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Imipenem/Cilastatin/XNW4107 (Experimental): Imipenem/Cilastatin 500mg/500mg in combination with XNW4107 250mg, Q6h (0.5h Infusion)
  Interventions: Drug: Combination of Imipenem/Cilastatin and XNW4107
- Imipenem/Cilastatin/Relebactam (Active Comparator): Imipenem/Cilastatin/Relebactam 1.25g Q6h (0.5h Infusion)
  Interventions: Drug: Imipenem/Cilastatin/Relebactam

INTERVENTIONS:
Drug: Combination of Imipenem/Cilastatin and XNW4107 — Imipenem/Cilastatin 500mg/500mg and XNW4107 250mg for Injection
  Arms: Imipenem/Cilastatin/XNW4107
Drug: Imipenem/Cilastatin/Relebactam — Imipenem/Cilastatin/Relebactam 1.25 g for Injection
  Other Names: Recarbrio
  Arms: Imipenem/Cilastatin/Relebactam

SUMMARY:
This study aims to compare treatment with Imipenem/Cilastatin-XNW4107 (IMI-XNW4107) with imipenem/cilastatin/relebactam (IMI/REL) in participants with hospital-acquired or ventilator-associated bacterial pneumonia (HABP or VAPB, respectively). The primary hypothesis is that IMI-XNW4107 is non-inferior to IMI/REL in all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Has HABP or VABP as defined below and requires treatment with IV antibiotic therapy. Fulfills clinical criteria, with onset of criteria occurring after more than 48 hours of hospitalization or within 7 days after discharge from a hospital (for HABP); or at least 48 hours after mechanical ventilation (for VABP)
2. Fulfills clinical criteria with symptoms or signs of cough, expectorated sputum production, dyspnea, worsening oxygenation, increase in respiratory secretions, fever/ hypothermia..
3. Fulfills laboratory test criteria with Leukocytosis/ Leukocytosis/ increase in immature neutrophils
4. Fulfill radiograph criteria with presence of new or progressive infiltrate(s) suggestive of bacterial pneumonia in X-ray/ Chest CT.
5. Female subjects of childbearing potential, who are willing to birth control during the study and for at least 30 days following the last dose of study medication. Male subjects with female sexual partners of childbearing potential are eligible for inclusion if they agree to use birth control for 90 days following the last dose of study medication. Male subjects must agree not to donate sperm

Exclusion Criteria:

1. Gram stain from a respiratory sample shows only Gram-positive cocci.
2. Have known or suspected community-acquired bacterial pneumonia, atypical pneumonia, viral pneumonia including Coronavirus disease, or chemical pneumonia.
3. Have HABP/VABP caused by an obstructive process, including lung cancer or other known obstruction.
4. Have received effective antibacterial drug therapy for the index infection of HABP/VABP for more than 24 hours during the previous 72 hours .
5. Have central nervous system infection.
6. Documented presence of immunodeficiency or an immunocompromised condition
7. Documented or severe hypersensitivity or previous severe adverse drug reaction, especially to any beta-lactam antibiotics, or any of the excipients used in the study drug formulations.
8. History of a seizure disorder requiring ongoing treatment with anti-convulsive therapy or prior treatment with anti-convulsive therapy within the last 3 years.
9. eGFR <15 mL/min/1.73㎡.
10. Patient is receiving hemodialysis or peritoneal dialysis.
11. Anticipated to be treated with any of Valproic acid or divalproex sodium, concomitant systemic Gram-negative antibacterial agents, or concomitant systemic antifungal or antiviral therapy for the index infection of HABP/VABP.
12. Life expectancy is <3 days.
13. Patients in refractory septic shock
14. Patients with 1 or more of laboratory abnormalities in baseline specimens.
15. History of active liver disease or cirrhosis.
16. APACHE II score of >30.
17. A female who is pregnant or breastfeeding or has a positive pregnancy test at Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2022-07-31 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2024-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Le, Study Chair — Evopoint Biosciences USA, Inc.)
Locations (35):
- United States (10):
  - Denver Health and Hospital Authority, Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Jackson Memorial Hospital (JMH) - Ryder Trauma Center, Miami, Florida
  - USF-TGH, Tampa, Florida
  - University of Maryland Medical Center, Baltimore, Maryland
  - Cox Health, Springfield, Missouri
  - VA medical center, Buffalo, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The University of Tennessee Medical Center, Knoxville, Tennessee
- France (11):
  - CHU de Nice, Nice, Alpes Maritimes
  - Hôpitaux Universitaires de Strasbourg, Strasbourg, Alsace
  - Nouvel Hopital CIVIL/ Medecine Intensive Reanimation, Strasbourg, Bas-Rhin
  - Chu Nimes, Nîmes, GARD
  - Chu Reims- Medical Icu, Reims, Grand Est
  - Cochin, Paris, Paris
  - Groupe Hospitalier Paris Saint-Joseph, Paris, Paris
  - APHP, Paris, Paris
  - intensive Unit Care CHU Amiens Picardie, Amiens, Picardie
  - CH victor dupouy, Argenteuil
  - Hôpital Foch, Suresnes, Île-de-France Region
- Israel (8):
  - Sheba Medical Center, Ramat Gan, Center
  - Wolfson Medical Center, H̱olon, Central District
  - Bnei-Zion Medical Center, Haifa, Haifa District
  - Shamir Medical Center, Be’er Ya‘aqov, HaMercaz
  - Hillel Yaffe Medical Center, Hadera, Israel
  - Rambam Critical Care division, Haifa, Israel
  - Tel Aviv Medical Center, Tel Aviv, Israel
  - Galilee Medical Center / Department int med A, Nahariya, Western Galilee
- Spain (6):
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Universitari Vall Hebron, Barcelona, Barcelona
  - Hospital Clínic of Barcelona, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Bellvitge University Hospital, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Tarragona Joan XXIII, Tarragona, Tarragona

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with a clinical diagnosis of hospital-acquired bacterial pneumonia (HABP)/ventilator-associated bacterial pneumonia (VABP) who met all eligibility criteria, and were assessed by the investigator as requiring 7 up to 14 days of intravenous (IV) antibiotic treatment in the hospital were randomized.
Groups:
- Imipenem/Cilastatin and XNW4107: Participants received imipenem/cilastatin via IV infusion and XNW4107 via injection during the treatment period of up to 14 days.
- Imipenem/Cilastatin/Relebactam: Participants received imipenem/cilastatin/relebactam via IV infusion during the treatment period of up to 14 days.
Period: Overall Study
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Started | 300 | 150
Received at Least 1 Dose | 299 | 150
Completed | 261 | 139
Not Completed | 39 | 11
Not completed — Other than Specified | 2 | 1
Not completed — Death | 18 | 4
Not completed — Lost to Follow-up | 6 | 3
Not completed — Withdrawal by Subject | 12 | 3
Not completed — Enrolled, Not Treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Measured in the Intention-to-Treat population, which included all participants who were randomized.
Groups:
- Imipenem/Cilastatin and XNW4107: Participants received imipenem/cilastatin via intravenous (IV) infusion and XNW4107 via injection during the treatment period of up to 14 days.
- Total: Total of all reporting groups
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam | Total
Number analyzed (Participants) | 300 | 150 | 450
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0
  Adults (18-64 years) | 168 | 86 | 254
  From 65-84 years | 121 | 61 | 182
  85 years and over | 11 | 3 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 50 | 136
  Male | 214 | 100 | 314
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 300 | 150 | 450
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 296 | 149 | 445
  White | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Day 14 All-cause Mortality Rate
Description: The all-cause mortality rate at Day 14 was calculated as the percentage of participants in each treatment group who experienced mortality, regardless of the cause, from randomization up to Day 14.
Time Frame: Day 14
Population: Measured in the Modified Intent-To-Treat (MITT) population, which included all participants from the Intent-to-Treat (ITT) who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 299 | 150
percentage of participants | 3.0 | 2.7
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Test type: Other; Treatment difference = 0.2, 95% CI 2-sided [-3.5 to 4.0]

2. Secondary Outcome: Day 28 All-cause Mortality Rate
Description: The all-cause mortality rate at Day 28 was calculated as the percentage of participants in each treatment group who experienced mortality, regardless of the cause, from randomization up to Day 28.
Time Frame: Day 28
Population: Measured in the MITT, which included all participants from the ITT who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 299 | 150
percentage of participants | 7.7 | 3.3
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Test type: Other; Treatment difference = 4.1, 95% CI 2-sided [-0.4 to 8.7]

3. Secondary Outcome: Day 14 and Day 28 All-cause Mortality Rate in the Micro-MITT Population
Description: The all-cause mortality rate at Day 14 and Day 28 was calculated as the percentage of participants in each treatment group who experienced mortality, regardless of the cause, from randomization up to Day 14 and Day 28.
Time Frame: Day 14, Day 28
Population: Measured in the microbiologic (micro)-MITT population, which included all participants from the MITT who had a Gram-negative pathogen identified at baseline and the pathogen was susceptible to the investigational medicinal product and comparator.
Measure: Number; unit: percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 113 | 57
percentage of participants
  Day 14 | 3.5 | 0
  Day 28 | 6.2 | 1.8
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Day 14; Test type: Other; Treatment difference = 3.2, 95% CI 2-sided [-3.0 to 9.4]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Day 28; Test type: Other; Treatment difference = 4.0, 95% CI 2-sided [-3.4 to 11.3]

4. Secondary Outcome: Day 14 and Day 28 All-cause Mortality Rate in the Extended Micro-MITT
Description: as for outcome 3
Time Frame: Day 14, Day 28
Population: Measured in the Extended micro-MITT population, which included all participants from the MITT who had a baseline Gram-negative pathogen identified which was susceptible to either the investigational medicinal product or comparator.
Measure: Number; unit: percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 153 | 78
percentage of participants
  Day 14 | 3.3 | 2.6
  Day 28 | 7.2 | 3.8
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Day 14; Test type: Other; Treatment difference = 0.5, 95% CI 2-sided [-5.4 to 6.3]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Day 28; Test type: Other; Treatment difference = 2.9, 95% CI 2-sided [-3.9 to 9.8]

5. Secondary Outcome: Day 14 and Day 28 All-cause Mortality Rate in the Clinically Evaluable (CE) Population
Description: as for outcome 3
Time Frame: Day 14, Day 28
Population: Measured in the CE population, which included all participants from the MITT who received at least 72 hours of IV study treatment, had an appropriate diagnosis of hospital-acquired bacterial pneumonia (HABP)/ventilator-associated bacterial pneumonia (VABP), had no important protocol deviations that affected the assessment of clinical outcome, and had no missing nor indeterminate assessment of clinical outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 233 | 120
percentage of participants
  Day 14 | 1.7 | 2.5
  Day 28 | 5.6 | 3.3
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Day 14; Test type: Other; Treatment difference = -0.8, 95% CI 2-sided [-4.9 to 3.3]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Day 28; Test type: Other; Treatment difference = 2.2, 95% CI 2-sided [-2.7 to 7.2]

6. Secondary Outcome: Day 14 and Day 28 All-cause Mortality Rate in the Microbiologically Evaluable (ME) Population
Description: as for outcome 3
Time Frame: Day 14, Day 28
Population: Measured in the ME population, which included all participants from the micro-MITT who received at least 72 hours of IV study treatment, had an appropriate diagnosis of HABP/VABP, had no important protocol deviations that affected the assessment of microbiological outcome, and had no missing nor indeterminate assessment of microbiological outcome. 'n' = participants evaluable at specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 96 | 51
percentage of participants
  Day 14 | 2.1 | 0
  Day 28 | 3.1 | 2.0
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Day 14; Test type: Other; Treatment difference = 2.1, 95% CI 2-sided [-4.7 to 8.9]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Day 28; Test type: Other; Treatment difference = 1.3, 95% CI 2-sided [-6.5 to 9.1]

7. Secondary Outcome: Day 14 and Day 28 All-cause Mortality Rate in the Carbapenem-resistant MITT (CR-MITT) Population
Description: as for outcome 3
Time Frame: Day 14, Day 28
Population: Measured in the CR-MITT Population, which included all participants from the MITT who had a baseline Gram-negative pathogen identified which is resistant to any carbapenem.
Measure: Number; unit: percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 53 | 23
percentage of participants
  Day 14 | 1.9 | 8.7
  Day 28 | 1.9 | 8.7
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Day 14; Test type: Other; Treatment difference = -7.8, 95% CI 2-sided [-25.3 to 9.7]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Day 28; Test type: Other; Treatment difference = -7.8, 95% CI 2-sided [-25.3 to 9.7]

8. Secondary Outcome: The Percentage of Participants With Clinical Success as Evaluated by the Investigator in the MITT Population
Description: Clinical success was defined as: For Day 4 visit: a participant was alive with resolution or improvement in at least 1 baseline sign/symptom AND no worsening of any baseline signs/symptoms AND no development of new signs/symptoms of pneumonia requiring the initiation of a non-study antibacterial therapy for the index infection. For end of treatment (EOT) or test-of-cure (TOC) visits: a participant was alive with complete resolution or significant improvement of signs and symptoms that were present at baseline and no new signs/symptoms of pneumonia, such that no further antibacterial therapy is necessary. For LFU, Clinical success at TOC with sustained resolution or marked improvement of baseline signs and symptoms of pneumonia during TOC and LFU without antimicrobial therapy (pneumonia).
Time Frame: Day 4, end of treatment (EOT) (up to Day 14), Test-of-Cure (TOC) (Day 21), and Late Follow-up (LFU) (Day 28)
Population: Measured in the MITT, which included all participants from the ITT who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 299 | 150
percentage of participants
  Day 4 | 59.2 | 56.0
  EOT (up to Day 14) | 74.6 | 71.3
  TOC (Day 21) | 62.9 | 63.3
  LFU (Day 28) | 58.9 | 56.7
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Day 4; Test type: Other; Treatment difference = 3.6, 95% CI 2-sided [-6.0 to 13.2]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; EOT (up to Day 14); Test type: Other; Treatment difference = 3.5, 95% CI 2-sided [-5.3 to 12.3]
Statistical Analysis 3: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; TOC (Day 21); Test type: Other; Treatment difference = -0.0, 95% CI 2-sided [-9.4 to 9.3]
Statistical Analysis 4: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; LFU (Day 28); Test type: Other; Treatment difference = 2.7, 95% CI 2-sided [-6.9 to 12.2]

9. Secondary Outcome: The Percentage of Participants With Clinical Success as Evaluated by the Investigator in the Micro-MITT Population
Description: Clinical success was defined as: For Day 4 visit: a participant was alive with resolution or improvement in at least 1 baseline sign/symptom AND no worsening of any baseline signs/symptoms AND no development of new signs/symptoms of pneumonia requiring the initiation of a non-study antibacterial therapy for the index infection. For EOT or TOC visits: a participant was alive with complete resolution or significant improvement of signs and symptoms that were present at baseline and no new signs/symptoms of pneumonia, such that no further antibacterial therapy is necessary. For LFU, Clinical success at TOC with sustained resolution or marked improvement of baseline signs and symptoms of pneumonia during TOC and LFU without antimicrobial therapy (pneumonia).
Time Frame: Day 4, EOT (up to Day 14), TOC (Day 21), and LFU (Day 28)
Population: Measured in the micro-MITT, which included all participants from the MITT who had a Gram-negative pathogen identified at baseline and the pathogen was susceptible to the investigational medicinal product and comparator.
Measure: Number; unit: percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 113 | 57
percentage of participants
  Day 4 | 54.0 | 56.1
  EOT (up to Day 14) | 84.1 | 71.9
  TOC (Day 21) | 66.4 | 61.4
  LFU (Day 28) | 62.8 | 54.4
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Day 4; Test type: Other; Treatment difference = -2.2, 95% CI 2-sided [-18.1 to 13.6]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; EOT (up to Day 14); Test type: Other; Treatment difference = 12.3, 95% CI 2-sided [-1.6 to 26.3]
Statistical Analysis 3: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; TOC (Day 21); Test type: Other; Treatment difference = 5.0, 95% CI 2-sided [-10.5 to 20.4]
Statistical Analysis 4: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; LFU (Day 28); Test type: Other; Treatment difference = 8.9, 95% CI 2-sided [-6.9 to 24.7]

10. Secondary Outcome: The Percentage of Participants With Clinical Success as Evaluated by the Investigator in the Extended Micro-MITT
Description: as for outcome 9
Time Frame: Day 4, EOT (up to Day 14), TOC (Day 21), and LFU (Day 28)
Population: Measured in the Extended micro-MITT, which included all participants from the MITT who had a baseline Gram-negative pathogen identified which was susceptible to either the investigational medicinal product or comparator.
Measure: Number; unit: percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 153 | 78
percentage of participants
  Day 4 | 56.2 | 56.4
  EOT (up to Day 14) | 81.0 | 73.1
  TOC (Day 21) | 65.4 | 57.7
  LFU (Day 28) | 60.8 | 51.3
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Day 4; Test type: Other; Treatment difference = 0.8, 95% CI 2-sided [-12.7 to 14.4]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; EOT (up to Day 14); Test type: Other; Treatment difference = 8.3, 95% CI 2-sided [-3.7 to 20.3]
Statistical Analysis 3: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; TOC (Day 21); Test type: Other; Treatment difference = 8.6, 95% CI 2-sided [-4.8 to 21.9]
Statistical Analysis 4: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; LFU (Day 28); Test type: Other; Treatment difference = 10.6, 95% CI 2-sided [-3.0 to 24.2]

11. Secondary Outcome: The Percentage of Participants With Clinical Success as Evaluated by the Investigator in the CE Population
Description: as for outcome 9
Time Frame: Day 4, end of treatment (EOT) (up to Day 14), Test-of-Cure (TOC) (Day 21), and Late Follow-up (LFU) (Day 28)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 233 | 120
percentage of participants
  Day 4 | 65.7 | 63.3
  EOT (up to Day 14) | 85.0 | 83.3
  TOC (Day 21) | 75.5 | 75.0
  LFU (Day 28) | 70.8 | 68.3
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Day 4; Test type: Other; Treatment difference = 2.3, 95% CI 2-sided [-8.3 to 12.8]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; EOT (up to Day 14); Test type: Other; Treatment difference = 1.7, 95% CI 2-sided [-6.7 to 10.1]
Statistical Analysis 3: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; TOC (Day 21); Test type: Other; Treatment Difference = 0.4, 95% CI 2-sided [-9.2 to 10.0]
Statistical Analysis 4: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; LFU (Day 28); Test type: Other; Treatment difference = 2.5, 95% CI 2-sided [-7.7 to 12.6]

12. Secondary Outcome: The Percentage of Participants With Clinical Success as Evaluated by the Investigator in the ME Population
Description: as for outcome 9
Time Frame: Day 4, end of treatment (EOT) (up to Day 14), Test-of-Cure (TOC) (Day 21), and Late Follow-up (LFU) (Day 28)
Population: Measured in the ME population, which included all participants from the micro-MITT who received at least 72 hours of IV study treatment, had an appropriate diagnosis of HABP/VABP, had no important protocol deviations that affected the assessment of microbiological outcome, and had no missing nor indeterminate assessment of microbiological outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 96 | 51
Percentage of participants
  Day 4 | 57.3 | 60.8
  EOT (up to Day 14) | 88.5 | 80.4
  TOC (Day 21) | 76.0 | 68.6
  LFU (Day 28) | 71.9 | 60.8
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Day 4; Test type: Other; Treatment difference = -4.6, 95% CI 2-sided [-21.4 to 12.2]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; EOT (up to Day 14); Test type: Other; Treatment difference = 7.7, 95% CI 2-sided [-5.8 to 21.2]
Statistical Analysis 3: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; TOC (Day 21); Test type: Other; Treatment difference = 6.3, 95% CI 2-sided [-9.4 to 22.0]
Statistical Analysis 4: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; LFU (Day 28); Test type: Other; Treatment difference = 10.6, 95% CI 2-sided [-5.9 to 27.1]

13. Secondary Outcome: The Percentage of Participants With Clinical Success as Evaluated by the Investigator in the CR-MITT Population
Description: as for outcome 9
Time Frame: Day 4, end of treatment (EOT) (up to Day 14), Test-of-Cure (TOC) (Day 21), and Late Follow-up (LFU) (Day 28)
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 53 | 23
Percentage of participants
  Day 4 | 60.4 | 56.5
  EOT (up to Day 14) | 79.2 | 60.9
  TOC (Day 21) | 64.2 | 43.5
  LFU (Day 28) | 50.9 | 39.1
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Day 4; Test type: Other; Treatment difference = 5.9, 95% CI 2-sided [-20.3 to 32.1]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; EOT (up to Day 14); Test type: Other; Treatment difference = 18.3, 95% CI 2-sided [-5.4 to 42.1]
Statistical Analysis 3: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; TOC (Day 21); Test type: Other; Treatment difference = 23.0, 95% CI 2-sided [-1.5 to 47.5]
Statistical Analysis 4: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; LFU (Day 28); Test type: Other; Treatment difference = 14.0, 95% CI 2-sided [-11.6 to 39.7]

14. Secondary Outcome: The Percentage of Participants With Microbiological Success in the Micro-MITT Population
Description: Microbiological success was defined as: • Eradication: Absence of the baseline Gram-negative pathogen from an appropriate clinical specimen • Presumed eradication: Absence of appropriate post-baseline culture material in a participant, but judged to be a clinical success.
Time Frame: EOT (up to Day 14), TOC (Day 21), and LFU (Day 28)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 113 | 57
percentage of participants
  EOT (up to Day 14) | 81.4 | 70.2
  TOC (Day 21) | 57.5 | 50.9
  LFU (Day 28) | 52.2 | 43.9
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; EOT (up to Day 14); Test type: Other; Treatment difference = 10.9, 95% CI 2-sided [-3.5 to 25.3]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; TOC (Day 21); Test type: Other; Treatment difference = 6.3, 95% CI 2-sided [-9.7 to 22.4]
Statistical Analysis 3: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; LFU (Day 28); Test type: Other; Treatment difference = 8.7, 95% CI 2-sided [-7.3 to 24.7]

15. Secondary Outcome: The Percentage of Participants With Microbiological Success in the Extended Micro-MITT Population
Description: as for outcome 14
Time Frame: EOT (up to Day 14), TOC (Day 21), and LFU (Day 28)
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 153 | 78
Percentage of participants
  EOT (up to Day 14) | 75.8 | 65.4
  TOC (Day 21) | 52.9 | 47.4
  LFU (Day 28) | 46.4 | 42.3
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; EOT (up to Day 14); Test type: Other; Treatment difference = 10.6, 95% CI 2-sided [-2.3 to 23.5]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; TOC (Day 21); Test type: Other; Treatment difference = 6.4, 95% CI 2-sided [-7.2 to 20.0]
Statistical Analysis 3: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; LFU (Day 28); Test type: Other; Treatment difference = 5.3, 95% CI 2-sided [-8.2 to 18.9]

16. Secondary Outcome: The Percentage of Participants With Microbiological Success in the CR-MITT Population
Description: as for outcome 14
Time Frame: EOT (up to Day 14), TOC (Day 21), and LFU (Day 28)
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 53 | 23
Percentage of participants
  EOT (up to Day 14) | 56.6 | 34.8
  TOC (Day 21) | 28.3 | 26.1
  LFU (Day 28) | 17.0 | 26.1
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; EOT (up to Day 14); Test type: Other; Treatment difference = 19.2, 95% CI 2-sided [-6.4 to 44.8]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; TOC (Day 21); Test type: Other; Treatment difference = -1.2, 95% CI 2-sided [-24.3 to 22.0]
Statistical Analysis 3: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; LFU (Day 28); Test type: Other; Treatment difference = -10.2, 95% CI 2-sided [-32.9 to 12.5]

17. Secondary Outcome: The Percentage of Participants With Microbiological Success in the ME Population
Description: as for outcome 14
Time Frame: EOT (up to Day 14), TOC (Day 21), and LFU (Day 28)
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 96 | 51
Percentage of participants
  EOT (up to Day 14) | 85.4 | 78.4
  TOC (Day 21) | 65.6 | 56.9
  LFU (Day 28) | 58.3 | 49.0
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; EOT (up to Day 14); Test type: Other; Treatment difference = 6.3, 95% CI 2-sided [-7.9 to 20.4]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; TOC (Day 21); Test type: Other; Treatment difference = 7.5, 95% CI 2-sided [-9.5 to 24.5]
Statistical Analysis 3: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; LFU (Day 28); Test type: Other; Treatment difference = 8.7, 95% CI 2-sided [-8.6 to 26.0]

18. Secondary Outcome: The Percentage of Participants With Microbiological Success by Pathogen in the Micro-MITT Population
Description: as for outcome 14
Time Frame: EOT (up to Day 14), TOC (Day 21), and LFU (Day 28)
Population: Measured in the micro-MITT, which included all participants from the MITT who had a Gram-negative pathogen identified at baseline and the pathogen was susceptible to the investigational medicinal product and comparator. Overall number of participants analysed=participants evaluable for the endpoint, n=number evaluable at the specified timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 76 | 37
Percentage of participants
  K.pneumoniae complex EOT (up to Day 14) | 88.2 | 64.9
  K.pneumoniae complex TOC (Day 21) | 61.8 | 54.1
  K.pneumoniae complex LFU (Day 28) | 57.9 | 45.9
  Pseudomonas aeruginosa EOT (up to Day 14): number analyzed (Participants) | 25 | 11
  Pseudomonas aeruginosa EOT (up to Day 14) | 68.0 | 45.5
  Pseudomonas aeruginosa TOC (Day 21): number analyzed (Participants) | 25 | 11
  Pseudomonas aeruginosa TOC (Day 21) | 36.0 | 27.3
  Pseudomonas aeruginosa LFU (Day 28): number analyzed (Participants) | 25 | 11
  Pseudomonas aeruginosa LFU (Day 28) | 28.0 | 27.3
  A.calco/baumannii complex EOT (up to Day 14): number analyzed (Participants) | 11 | 11
  A.calco/baumannii complex EOT (up to Day 14) | 72.7 | 72.7
  A.calco/baumannii complex TOC (Day 21): number analyzed (Participants) | 11 | 11
  A.calco/baumannii complex TOC (Day 21) | 72.7 | 72.7
  A.calco/baumannii complex LFU (Day 28): number analyzed (Participants) | 11 | 11
  A.calco/baumannii complex LFU (Day 28) | 72.7 | 63.6
  Enterobacter cloacae complex EOT (up to Day 14): number analyzed (Participants) | 5 | 2
  Enterobacter cloacae complex EOT (up to Day 14) | 60.0 | 100.0
  Enterobacter cloacae complex TOC (Day 21): number analyzed (Participants) | 5 | 2
  Enterobacter cloacae complex TOC (Day 21) | 40.0 | 100.0
  Enterobacter cloacae complex LFU (Day 28): number analyzed (Participants) | 5 | 2
  Enterobacter cloacae complex LFU (Day 28) | 40.0 | 100.0
  Klebsiella aerogenes EOT (up to Day 14): number analyzed (Participants) | 3 | 3
  Klebsiella aerogenes EOT (up to Day 14) | 66.7 | 100.0
  Klebsiella aerogenes TOC (Day 21): number analyzed (Participants) | 3 | 3
  Klebsiella aerogenes TOC (Day 21) | 33.3 | 33.3
  Klebsiella aerogenes LFU (Day 28): number analyzed (Participants) | 3 | 3
  Klebsiella aerogenes LFU (Day 28) | 33.3 | 33.3
  Escherichia coli EOT (up to Day 14): number analyzed (Participants) | 3 | 1
  Escherichia coli EOT (up to Day 14) | 100.0 | 100.0
  Escherichia coli TOC (Day 21): number analyzed (Participants) | 3 | 1
  Escherichia coli TOC (Day 21) | 66.7 | 100.0
  Escherichia coli LFU (Day 28): number analyzed (Participants) | 3 | 1
  Escherichia coli LFU (Day 28) | 66.7 | 100.0
  Citrobacter koseri EOT (up to Day 14): number analyzed (Participants) | 1 | 2
  Citrobacter koseri EOT (up to Day 14) | 100.0 | 100.0
  Citrobacter koseri TOC (Day 21): number analyzed (Participants) | 1 | 2
  Citrobacter koseri TOC (Day 21) | 100.0 | 50.0
  Citrobacter koseri LFU (Day 28): number analyzed (Participants) | 1 | 2
  Citrobacter koseri LFU (Day 28) | 0.0 | 50.0
  Acinetobacter junii EOT (up to Day 14): number analyzed (Participants) | 1 | 1
  Acinetobacter junii EOT (up to Day 14) | 100.0 | 100.0
  Acinetobacter junii TOC (Day 21): number analyzed (Participants) | 1 | 1
  Acinetobacter junii TOC (Day 21) | 100.0 | 100.0
  Acinetobacter junii LFU (Day 28): number analyzed (Participants) | 1 | 1
  Acinetobacter junii LFU (Day 28) | 100.0 | 100.0
  Klebsiella oxytoca EOT (up to Day 14): number analyzed (Participants) | 1 | 1
  Klebsiella oxytoca EOT (up to Day 14) | 100.0 | 100.0
  Klebsiella oxytoca TOC (Day 21): number analyzed (Participants) | 1 | 1
  Klebsiella oxytoca TOC (Day 21) | 0.0 | 100.0
  Klebsiella oxytoca LFU (Day 28): number analyzed (Participants) | 1 | 1
  Klebsiella oxytoca LFU (Day 28) | 0.0 | 100.0
  Citrobacter freundii complex EOT (up to Day 14): number analyzed (Participants) | 1 | 0
  Citrobacter freundii complex EOT (up to Day 14) | 100.0 |
  Citrobacter freundii complex TOC (Day 21): number analyzed (Participants) | 1 | 0
  Citrobacter freundii complex TOC (Day 21) | 100.0 |
  Citrobacter freundii complex LFU (Day 28): number analyzed (Participants) | 1 | 0
  Citrobacter freundii complex LFU (Day 28) | 100.0 |
  Serratia marcescens EOT (up to Day 14): number analyzed (Participants) | 0 | 1
  Serratia marcescens EOT (up to Day 14) |  | 0.0
  Serratia marcescens TOC (Day 21): number analyzed (Participants) | 0 | 1
  Serratia marcescens TOC (Day 21) |  | 100.0
  Serratia marcescens LFU (Day 28): number analyzed (Participants) | 0 | 1
  Serratia marcescens LFU (Day 28) |  | 0.0
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella pneumoniae complex EOT (up to Day 14); Test type: Other; Treatment difference = 23.3, 95% CI 2-sided [4.3 to 42.3]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella pneumoniae complex TOC (Day 21); Test type: Other; Treatment difference = 7.8, 95% CI 2-sided [-13.6 to 29.2]
Statistical Analysis 3: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella pneumoniae complex LFU (Day 28); Test type: Other; Treatment difference = 11.9, 95% CI 2-sided [-9.6 to 33.5]
Statistical Analysis 4: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Pseudomonas aeruginosa EOT (up to Day 14); Test type: Other; Treatment difference = 22.5, 95% CI 2-sided [-18.6 to 63.7]
Statistical Analysis 5: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Pseudomonas aeruginosa TOC (Day 21); Test type: Other; Treatment difference = 8.7, 95% CI 2-sided [-30.2 to 47.6]
Statistical Analysis 6: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Pseudomonas aeruginosa LFU (Day 28); Test type: Other; Treatment difference = 0.7, 95% CI 2-sided [-37.5 to 38.9]
Statistical Analysis 7: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; A.calco/baumannii complex EOT (up to Day 14); Test type: Other; Treatment difference = 0.0, 95% CI 2-sided [-46.3 to 46.3]
Statistical Analysis 8: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; A.calco/baumannii complex TOC (Day 21); Test type: Other; Treatment difference = 0.0, 95% CI 2-sided [-46.3 to 46.3]
Statistical Analysis 9: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; A.calco/baumannii complex LFU (Day 28); Test type: Other; Treatment difference = 9.1, 95% CI 2-sided [-38.7 to 56.9]
Statistical Analysis 10: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Enterobacter cloacae complex EOT (up to Day 14); Test type: Other; Treatment difference = -40.0, 95% CI 2-sided [-100.0 to 37.9]
Statistical Analysis 11: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Enterobacter cloacae complex TOC (Day 21); Test type: Other; Treatment difference = -60.0, 95% CI 2-sided [-100.0 to 17.9]
Statistical Analysis 12: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Enterobacter cloacae complex LFU (Day 28); Test type: Other; Treatment difference = -60.0, 95% CI 2-sided [-100.0 to 17.9]
Statistical Analysis 13: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella aerogenes EOT (up to Day 14); Test type: Other; Treatment difference = -33.3, 95% CI 2-sided [-100.0 to 53.3]
Statistical Analysis 14: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella aerogenes TOC (Day 21); Test type: Other; Treatment difference = 0.0, 95% CI 2-sided [-100.0 to 100.0]
Statistical Analysis 15: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella aerogenes LFU (Day 28); Test type: Other; Treatment difference = 0.0, 95% CI 2-sided [-100.0 to 100.0]
Statistical Analysis 16: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Escherichia coli TOC (Day 21); Test type: Other; Treatment difference = -33.3, 95% CI 2-sided [-100.0 to 86.7]
Statistical Analysis 17: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Escherichia coli LFU (Day 28); Test type: Other; Treatment difference = -33.3, 95% CI 2-sided [-100.0 to 86.7]
Statistical Analysis 18: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Citrobacter koseri TOC (Day 21); Test type: Other; Treatment difference = 50.0, 95% CI 2-sided [-94.3 to 100.0]
Statistical Analysis 19: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Citrobacter koseri LFU (Day 28); Test type: Other; Treatment difference = -50.0, 95% CI 2-sided [-100.0 to 94.3]
Statistical Analysis 20: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella oxytoca TOC (Day 21); Test type: Other; Treatment difference = -100.0, 95% CI 2-sided [-100.0 to 0.0]
Statistical Analysis 21: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella oxytoca LFU (Day 28); Test type: Other; Treatment difference = -100.0, 95% CI 2-sided [-100.0 to 0.0]

19. Secondary Outcome: The Percentage of Participants With Microbiological Success by Pathogen in the Extended Micro-MITT Population
Description: as for outcome 14
Time Frame: EOT (up to Day 14), TOC (Day 21), and LFU (Day 28)
Population: Measured in the Extended micro-MITT, which included all participants from the MITT who had a baseline Gram-negative pathogen identified which was susceptible to either the investigational medicinal product or comparator. Overall number of participants analysed=participants evaluable for the endpoint, n=number evaluable at the specified timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 89 | 43
Percentage of participants
  K.pneumoniae complex EOT (up to Day 14) | 85.4 | 67.4
  K.pneumoniae complex TOC (Day 21) | 58.4 | 58.1
  K.pneumoniae complex LFU (Day 28) | 53.9 | 51.2
  A.calco/baumannii complex EOT (up to Day 14): number analyzed (Participants) | 28 | 23
  A.calco/baumannii complex EOT (up to Day 14) | 75.0 | 56.5
  A.calco/baumannii complex TOC (Day 21): number analyzed (Participants) | 28 | 23
  A.calco/baumannii complex TOC (Day 21) | 57.1 | 47.8
  A.calco/baumannii complex LFU (Day 28): number analyzed (Participants) | 28 | 23
  A.calco/baumannii complex LFU (Day 28) | 46.4 | 43.5
  Pseudomonas aeruginosa EOT (up to Day 14): number analyzed (Participants) | 32 | 14
  Pseudomonas aeruginosa EOT (up to Day 14) | 59.4 | 50.0
  Pseudomonas aeruginosa TOC (Day 21): number analyzed (Participants) | 32 | 14
  Pseudomonas aeruginosa TOC (Day 21) | 34.4 | 28.6
  Pseudomonas aeruginosa LFU (Day 28): number analyzed (Participants) | 32 | 14
  Pseudomonas aeruginosa LFU (Day 28) | 28.1 | 28.6
  Burkholderia cepacia complex EOT (up to Day 14): number analyzed (Participants) | 6 | 3
  Burkholderia cepacia complex EOT (up to Day 14) | 66.7 | 100.0
  Burkholderia cepacia complex TOC (Day 21): number analyzed (Participants) | 6 | 3
  Burkholderia cepacia complex TOC (Day 21) | 66.7 | 66.7
  Burkholderia cepacia complex LFU (Day 28): number analyzed (Participants) | 6 | 3
  Burkholderia cepacia complex LFU (Day 28) | 66.7 | 66.7
  Klebsiella aerogenes EOT (Up to Day 14): number analyzed (Participants) | 6 | 3
  Klebsiella aerogenes EOT (Up to Day 14) | 66.7 | 100.0
  Klebsiella aerogenes TOC (Day 21): number analyzed (Participants) | 6 | 3
  Klebsiella aerogenes TOC (Day 21) | 50.0 | 33.3
  Klebsiella aerogenes LFU (Day 28): number analyzed (Participants) | 6 | 3
  Klebsiella aerogenes LFU (Day 28) | 50.0 | 33.3
  Enterobacter cloacae complex EOT (up to Day 14): number analyzed (Participants) | 5 | 3
  Enterobacter cloacae complex EOT (up to Day 14) | 60.0 | 100.0
  Enterobacter cloacae complex TOC (Day 21): number analyzed (Participants) | 5 | 3
  Enterobacter cloacae complex TOC (Day 21) | 40.0 | 100.0
  Enterobacter cloacae complex LFU (Day 28): number analyzed (Participants) | 5 | 3
  Enterobacter cloacae complex LFU (Day 28) | 40.0 | 66.7
  Escherichia coli EOT (up to Day 14): number analyzed (Participants) | 4 | 2
  Escherichia coli EOT (up to Day 14) | 100.0 | 100.0
  Escherichia coli TOC (Day 21): number analyzed (Participants) | 4 | 2
  Escherichia coli TOC (Day 21) | 75.0 | 100.0
  Escherichia coli LFU (Day 28): number analyzed (Participants) | 4 | 2
  Escherichia coli LFU (Day 28) | 50.0 | 100.0
  Haemophilus influenzae EOT (up to Day 14): number analyzed (Participants) | 5 | 0
  Haemophilus influenzae EOT (up to Day 14) | 100.0 |
  Haemophilus influenzae TOC (Day 21): number analyzed (Participants) | 5 | 0
  Haemophilus influenzae TOC (Day 21) | 100.0 |
  Haemophilus influenzae LFU (Day 28): number analyzed (Participants) | 5 | 0
  Haemophilus influenzae LFU (Day 28) | 100.0 |
  Citrobacter koseri EOT (up to Day 14): number analyzed (Participants) | 1 | 2
  Citrobacter koseri EOT (up to Day 14) | 100.0 | 100.0
  Citrobacter koseri TOC (Day 21): number analyzed (Participants) | 1 | 2
  Citrobacter koseri TOC (Day 21) | 100.0 | 50.0
  Citrobacter koseri LFU (Day 28): number analyzed (Participants) | 1 | 2
  Citrobacter koseri LFU (Day 28) | 0.0 | 50.0
  Proteus mirabilis EOT (up to Day 14): number analyzed (Participants) | 1 | 2
  Proteus mirabilis EOT (up to Day 14) | 0.0 | 0.0
  Proteus mirabilis TOC (Day 21): number analyzed (Participants) | 1 | 2
  Proteus mirabilis TOC (Day 21) | 0.0 | 0.0
  Proteus mirabilis LFU (Day 28): number analyzed (Participants) | 1 | 2
  Proteus mirabilis LFU (Day 28) | 0.0 | 0.0
  Acinetobacter junii EOT (up to Day 14): number analyzed (Participants) | 1 | 1
  Acinetobacter junii EOT (up to Day 14) | 100.0 | 100.0
  Acinetobacter junii TOC (Day 21): number analyzed (Participants) | 1 | 1
  Acinetobacter junii TOC (Day 21) | 100.0 | 100.0
  Acinetobacter junii LFU (Day 28): number analyzed (Participants) | 1 | 1
  Acinetobacter junii LFU (Day 28) | 100.0 | 100.0
  Citrobacter freundii complex EOT (up to Day 14): number analyzed (Participants) | 2 | 0
  Citrobacter freundii complex EOT (up to Day 14) | 100.0 |
  Citrobacter freundii complex TOC (Day 21): number analyzed (Participants) | 2 | 0
  Citrobacter freundii complex TOC (Day 21) | 100.0 |
  Citrobacter freundii complex LFU (Day 28): number analyzed (Participants) | 2 | 0
  Citrobacter freundii complex LFU (Day 28) | 100.0 |
  Klebsiella oxytoca EOT (up to Day 14): number analyzed (Participants) | 1 | 1
  Klebsiella oxytoca EOT (up to Day 14) | 100.0 | 100.0
  Klebsiella oxytoca TOC (Day 21): number analyzed (Participants) | 1 | 1
  Klebsiella oxytoca TOC (Day 21) | 0.0 | 100.0
  Klebsiella oxytoca LFU (Day 28): number analyzed (Participants) | 1 | 1
  Klebsiella oxytoca LFU (Day 28) | 0.0 | 100.0
  Serratia marcescens EOT (up to Day 14): number analyzed (Participants) | 1 | 1
  Serratia marcescens EOT (up to Day 14) | 100.0 | 0.0
  Serratia marcescens TOC (Day 21): number analyzed (Participants) | 1 | 1
  Serratia marcescens TOC (Day 21) | 0.0 | 100.0
  Serratia marcescens LFU (Day 28): number analyzed (Participants) | 1 | 1
  Serratia marcescens LFU (Day 28) | 0.0 | 0.0
  Morganella morganii EOT (up to Day 14): number analyzed (Participants) | 1 | 0
  Morganella morganii EOT (up to Day 14) | 100.0 |
  Morganella morganii TOC (Day 21): number analyzed (Participants) | 1 | 0
  Morganella morganii TOC (Day 21) | 100.0 |
  Morganella morganii LFU (Day 28): number analyzed (Participants) | 1 | 0
  Morganella morganii LFU (Day 28) | 100.0 |
  Pseudomonas otitidis EOT (up to Day 14): number analyzed (Participants) | 1 | 0
  Pseudomonas otitidis EOT (up to Day 14) | 100.0 |
  Pseudomonas otitidis TOC (Day 21): number analyzed (Participants) | 1 | 0
  Pseudomonas otitidis TOC (Day 21) | 100.0 |
  Pseudomonas otitidis LFU (Day 28): number analyzed (Participants) | 1 | 0
  Pseudomonas otitidis LFU (Day 28) | 100.0 |
  Ralstonia pickettii EOT (up to Day 14): number analyzed (Participants) | 1 | 0
  Ralstonia pickettii EOT (up to Day 14) | 100.0 |
  Ralstonia pickettii TOC (Day 21): number analyzed (Participants) | 1 | 0
  Ralstonia pickettii TOC (Day 21) | 100.0 |
  Ralstonia pickettii LFU (Day 28): number analyzed (Participants) | 1 | 0
  Ralstonia pickettii LFU (Day 28) | 100.0 |
  Sphingomonas species EOT (up to Day 14): number analyzed (Participants) | 0 | 1
  Sphingomonas species EOT (up to Day 14) |  | 100.0
  Sphingomonas species TOC (Day 21): number analyzed (Participants) | 0 | 1
  Sphingomonas species TOC (Day 21) |  | 100.0
  Sphingomonas species LFU (Day 28): number analyzed (Participants) | 0 | 1
  Sphingomonas species LFU (Day 28) |  | 100.0
  Stenotrophomonas maltophilia EOT (up to Day 14): number analyzed (Participants) | 0 | 1
  Stenotrophomonas maltophilia EOT (up to Day 14) |  | 0.0
  Stenotrophomonas maltophilia TOC (Day 21): number analyzed (Participants) | 0 | 1
  Stenotrophomonas maltophilia TOC (Day 21) |  | 0.0
  Stenotrophomonas maltophilia LFU (Day 28): number analyzed (Participants) | 0 | 1
  Stenotrophomonas maltophilia LFU (Day 28) |  | 0.0
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella pneumoniae complex EOT (up to Day 14); Test type: Other; Treatment difference = 18.0, 95% CI 2-sided [0.4 to 35.5]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; A.calco/baumannii complex EOT (up to Day 14); Test type: Other; Treatment difference = 18.5, 95% CI 2-sided [-11.3 to 48.3]
Statistical Analysis 3: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Pseudomonas aeruginosa EOT (up to Day 14); Test type: Other; Treatment difference = 9.4, 95% CI 2-sided [-27.0 to 45.7]
Statistical Analysis 4: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Burkholderia cepacia complex EOT (up to Day 14); Test type: Other; Treatment difference = -33.3, 95% CI 2-sided [-96.1 to 29.4]
Statistical Analysis 5: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella aerogenes EOT (up to Day 14); Test type: Other; Treatment difference = -33.3, 95% CI 2-sided [-96.1 to 29.4]
Statistical Analysis 6: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Enterobacter cloacae complex EOT (up to Day 14); Test type: Other; Treatment difference = -40.0, 95% CI 2-sided [-100.0 to 29.6]
Statistical Analysis 7: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Serratia marcescens EOT (up to Day 14); Test type: Other; Treatment difference = 100.0, 95% CI 2-sided [0.0 to 100.0]
Statistical Analysis 8: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella pneumoniae complex TOC (Day 21); Test type: Other; Treatment difference = 0.3, 95% CI 2-sided [-19.4 to 20.0]
Statistical Analysis 9: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; A.calco/baumannii complex TOC (Day 21); Test type: Other; Treatment difference = 9.3, 95% CI 2-sided [-22.1 to 40.7]
Statistical Analysis 10: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Pseudomonas aeruginosa TOC (Day 21); Test type: Other; Treatment difference = 5.8, 95% CI 2-sided [-28.2 to 39.8]
Statistical Analysis 11: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Burkholderia cepacia complex TOC (Day 21); Test type: Other; Treatment difference = 0.0, 95% CI 2-sided [-90.3 to 90.3]
Statistical Analysis 12: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella aerogenes TOC (Day 21); Test type: Other; Treatment difference = 16.7, 95% CI 2-sided [-75.0 to 100.0]
Statistical Analysis 13: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Enterobacter cloacae complex TOC (Day 21); Test type: Other; Treatment difference = -60.0, 95% CI 2-sided [-100.0 to 9.6]
Statistical Analysis 14: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Escherichia coli TOC (Day 21); Test type: Other; Treatment difference = -25.0, 95% CI 2-sided [-100.0 to 54.9]
Statistical Analysis 15: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Citrobacter koseri TOC (Day 21); Test type: Other; Treatment difference = 50.0, 95% CI 2-sided [-94.3 to 100.0]
Statistical Analysis 16: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella oxytoca TOC (Day 21); Test type: Other; Treatment difference = -100.0, 95% CI 2-sided [-100.0 to 0.0]
Statistical Analysis 17: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Serratia marcescens TOC (Day 21); Test type: Other; Treatment difference = -100.0, 95% CI 2-sided [-100.0 to 0.0]
Statistical Analysis 18: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella pneumoniae complex LFU (Day 28); Test type: Other; Treatment difference = 2.8, 95% CI 2-sided [-17.1 to 22.7]
Statistical Analysis 19: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; A.calco/baumannii complex LFU (Day 28); Test type: Other; Treatment difference = 3.0, 95% CI 2-sided [-28.4 to 34.3]
Statistical Analysis 20: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Pseudomonas aeruginosa LFU (Day 28); Test type: Other; Treatment difference = -0.4, 95% CI 2-sided [-33.9 to 33.0]
Statistical Analysis 21: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Burkholderia cepacia complex LFU (Day 28); Test type: Other; Treatment difference = 0.0, 95% CI 2-sided [-90.3 to 90.3]
Statistical Analysis 22: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella aerogenes LFU (Day 28); Test type: Other; Treatment difference = 16.7, 95% CI 2-sided [-75.0 to 100.0]
Statistical Analysis 23: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Enterobacter cloacae complex LFU (Day 28); Test type: Other; Treatment difference = -26.7, 95% CI 2-sided [-100.0 to 68.5]
Statistical Analysis 24: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Escherichia coli LFU (Day 28); Test type: Other; Treatment difference = -50.0, 95% CI 2-sided [-100.0 to 36.5]
Statistical Analysis 25: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Citrobacter koseri LFU (Day 28); Test type: Other; Treatment difference = -50.0, 95% CI 2-sided [-100.0 to 94.3]
Statistical Analysis 26: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella oxytoca LFU (Day 28); Test type: Other; Treatment difference = -100.0, 95% CI 2-sided [-100.0 to 0.0]

20. Secondary Outcome: The Percentage of Participants With Microbiological Success by Pathogen in the ME Population
Description: as for outcome 14
Time Frame: EOT (up to Day 14), TOC (Day 21), and LFU (Day 28)
Population: Measured in the ME population, which included all participants from the micro-MITT who received at least 72 hours of IV study treatment, had an appropriate diagnosis of HABP/VABP, had no important protocol deviations that affected the assessment of microbiological outcome, and had no missing nor indeterminate assessment of microbiological outcome. Overall number of participants analysed=participants evaluable for the endpoint, n=number evaluable at the specified timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 64 | 33
Percentage of participants
  K.pneumoniae complex EOT (up to Day 14) | 93.8 | 72.7
  K.pneumoniae complex TOC (Day 21) | 70.3 | 60.6
  K.pneumoniae complex LFU (Day 28) | 64.1 | 51.5
  Pseudomonas aeruginosa EOT (up to Day 14): number analyzed (Participants) | 22 | 10
  Pseudomonas aeruginosa EOT (up to Day 14) | 68.2 | 50.0
  Pseudomonas aeruginosa TOC (Day 21): number analyzed (Participants) | 22 | 10
  Pseudomonas aeruginosa TOC (Day 21) | 40.9 | 30.0
  Pseudomonas aeruginosa LFU (Day 28): number analyzed (Participants) | 22 | 10
  Pseudomonas aeruginosa LFU (Day 28) | 31.8 | 30.0
  A.calco/baumannii complex EOT (up to Day 14): number analyzed (Participants) | 10 | 9
  A.calco/baumannii complex EOT (up to Day 14) | 80.0 | 88.9
  A.calco/baumannii complex TOC (Day 21): number analyzed (Participants) | 10 | 9
  A.calco/baumannii complex TOC (Day 21) | 80.0 | 88.9
  A.calco/baumannii complex LFU (Day 28): number analyzed (Participants) | 10 | 9
  A.calco/baumannii complex LFU (Day 28) | 80.0 | 77.8
  Klebsiella aerogenes EOT (up to Day 14): number analyzed (Participants) | 2 | 3
  Klebsiella aerogenes EOT (up to Day 14) | 50.0 | 100.0
  Klebsiella aerogenes TOC (Day 21): number analyzed (Participants) | 2 | 3
  Klebsiella aerogenes TOC (Day 21) | 50.0 | 33.3
  Klebsiella aerogenes LFU (Day 28): number analyzed (Participants) | 2 | 3
  Klebsiella aerogenes LFU (Day 28) | 50.0 | 33.3
  Enterobacter cloacae complex EOT (up to Day 14): number analyzed (Participants) | 2 | 2
  Enterobacter cloacae complex EOT (up to Day 14) | 50.0 | 100.0
  Enterobacter cloacae complex TOC (Day 21): number analyzed (Participants) | 2 | 2
  Enterobacter cloacae complex TOC (Day 21) | 50.0 | 100.0
  Enterobacter cloacae complex LFU (Day 28): number analyzed (Participants) | 2 | 2
  Enterobacter cloacae complex LFU (Day 28) | 50.0 | 100.0
  Escherichia coli EOT (up to Day 14): number analyzed (Participants) | 3 | 1
  Escherichia coli EOT (up to Day 14) | 100.0 | 100.0
  Escherichia coli TOC (Day 21): number analyzed (Participants) | 3 | 1
  Escherichia coli TOC (Day 21) | 66.7 | 100.0
  Escherichia coli LFU (Day 28): number analyzed (Participants) | 3 | 1
  Escherichia coli LFU (Day 28) | 66.7 | 100.0
  Citrobacter koseri EOT (up to Day 14): number analyzed (Participants) | 1 | 2
  Citrobacter koseri EOT (up to Day 14) | 100.0 | 100.0
  Citrobacter koseri TOC (Day 21): number analyzed (Participants) | 1 | 2
  Citrobacter koseri TOC (Day 21) | 100.0 | 50.0
  Citrobacter koseri LFU (Day 28): number analyzed (Participants) | 1 | 2
  Citrobacter koseri LFU (Day 28) | 0.0 | 50.0
  Acinetobacter junii EOT (up to Day 14): number analyzed (Participants) | 1 | 1
  Acinetobacter junii EOT (up to Day 14) | 100.0 | 100.0
  Acinetobacter junii TOC (Day 21): number analyzed (Participants) | 1 | 1
  Acinetobacter junii TOC (Day 21) | 100.0 | 100.0
  Acinetobacter junii LFU (Day 28): number analyzed (Participants) | 1 | 1
  Acinetobacter junii LFU (Day 28) | 100.0 | 100.0
  Klebsiella oxytoca EOT (up to Day 14): number analyzed (Participants) | 1 | 1
  Klebsiella oxytoca EOT (up to Day 14) | 100.0 | 100.0
  Klebsiella oxytoca TOC (Day 21): number analyzed (Participants) | 1 | 1
  Klebsiella oxytoca TOC (Day 21) | 0.0 | 100.0
  Klebsiella oxytoca LFU (Day 28): number analyzed (Participants) | 1 | 1
  Klebsiella oxytoca LFU (Day 28) | 0.0 | 100.0
  Citrobacter freundii complex EOT (up to Day 14): number analyzed (Participants) | 1 | 0
  Citrobacter freundii complex EOT (up to Day 14) | 100.0 |
  Citrobacter freundii complex TOC (Day 21): number analyzed (Participants) | 1 | 0
  Citrobacter freundii complex TOC (Day 21) | 100.0 |
  Citrobacter freundii complex LFU (Day 28): number analyzed (Participants) | 1 | 0
  Citrobacter freundii complex LFU (Day 28) | 100.0 |
  Serratia marcescens EOT (up to Day 14): number analyzed (Participants) | 0 | 1
  Serratia marcescens EOT (up to Day 14) |  | 0.0
  Serratia marcescens TOC (Day 21): number analyzed (Participants) | 0 | 1
  Serratia marcescens TOC (Day 21) |  | 100.0
  Serratia marcescens LFU (Day 28): number analyzed (Participants) | 0 | 1
  Serratia marcescens LFU (Day 28) |  | 0.0
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella pneumoniae complex EOT (up to Day 14); Test type: Other; Treatment difference = 21.0, 95% CI 2-sided [2.4 to 39.6]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Pseudomonas aeruginosa EOT (up to Day 14); Test type: Other; Treatment difference = 18.2, 95% CI 2-sided [-25.7 to 62.0]
Statistical Analysis 3: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; A.calco/baumannii complex EOT (up to Day 14); Test type: Other; Treatment difference = -8.9, 95% CI 2-sided [-51.6 to 33.9]
Statistical Analysis 4: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella aerogenes EOT (up to Day 14); Test type: Other; Treatment difference = -50.0, 95% CI 2-sided [-100.0 to 61.0]
Statistical Analysis 5: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Enterobacter cloacae complex EOT (up to Day 14); Test type: Other; Treatment difference = -50.0, 95% CI 2-sided [-100.0 to 69.3]
Statistical Analysis 6: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella pneumoniae complex TOC (Day 21); Test type: Other; Treatment difference = 9.7, 95% CI 2-sided [-12.7 to 32.1]
Statistical Analysis 7: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Pseudomonas aeruginosa TOC (Day 21); Test type: Other; Treatment difference = 10.9, 95% CI 2-sided [-31.4 to 53.2]
Statistical Analysis 8: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; A.calco/baumannii complex TOC (Day 21); Test type: Other; Treatment difference = -8.9, 95% CI 2-sided [-51.6 to 33.9]
Statistical Analysis 9: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella aerogenes TOC (Day 21); Test type: Other; Treatment difference = 16.7, 95% CI 2-sided [-100.0 to 100]
Statistical Analysis 10: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Enterobacter cloacae complex TOC (Day 21); Test type: Other; Treatment difference = -50.0, 95% CI 2-sided [-100.0 to 69.3]
Statistical Analysis 11: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Escherichia coli TOC (Day 21); Test type: Other; Treatment difference = -33.3, 95% CI 2-sided [-100.0 to 86.7]
Statistical Analysis 12: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Citrobacter koseri TOC (Day 21); Test type: Other; Treatment difference = 50.0, 95% CI 2-sided [-94.3 to 100.0]
Statistical Analysis 13: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella oxytoca TOC (Day 21); Test type: Other; Treatment difference = -100.0, 95% CI 2-sided [-100.0 to 0.0]
Statistical Analysis 14: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella pneumoniae complex LFU (Day 28); Test type: Other; Treatment difference = 12.5, 95% CI 2-sided [-10.5 to 35.6]
Statistical Analysis 15: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Pseudomonas aeruginosa LFU (Day 28); Test type: Other; Treatment difference = 1.8, 95% CI 2-sided [-39.9 to 43.5]
Statistical Analysis 16: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; A.calco/baumannii complex LFU (Day 28); Test type: Other; Treatment difference = 2.2, 95% CI 2-sided [-45.1 to 49.6]
Statistical Analysis 17: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella aerogenes LFU (Day 28); Test type: Other; Treatment difference = 16.7, 95% CI 2-sided [-100.0 to 100.0]
Statistical Analysis 18: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Enterobacter cloacae complex LFU (Day 28); Test type: Other; Treatment difference = -50.0, 95% CI 2-sided [-100.0 to 69.3]
Statistical Analysis 19: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Escherichia coli LFU (Day 28); Test type: Other; Treatment difference = -33.3, 95% CI 2-sided [-100.0 to 86.7]
Statistical Analysis 20: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Citrobacter koseri LFU (Day 28); Test type: Other; Treatment difference = -50.0, 95% CI 2-sided [-100.0 to 94.3]
Statistical Analysis 21: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella oxytoca LFU (Day 28); Test type: Other; Treatment difference = -100.0, 95% CI 2-sided [-100.0 to 0.0]

21. Secondary Outcome: The Percentage of Participants With Microbiological Success by Pathogen in the CR-MITT Population
Description: as for outcome 14
Time Frame: EOT (up to Day 14), TOC (Day 21), and LFU (Day 28)
Population: Measured in the CR-MITT Population, which included all participants from the MITT who had a baseline Gram-negative pathogen identified which is resistant to any carbapenem. Overall number of participants analysed=participants evaluable for the endpoint, n=number evaluable at the specified timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 26 | 16
Percentage of participants
  A.calco/baumannii complex EOT (up to Day 14) | 61.5 | 31.3
  A.calco/baumannii complex TOC (Day 21) | 30.8 | 18.8
  A.calco/baumannii complex LFU (Day 28) | 19.2 | 18.8
  Klebsiella pneumoniae complex EOT (up to Day 14): number analyzed (Participants) | 19 | 7
  Klebsiella pneumoniae complex EOT (up to Day 14) | 63.2 | 71.4
  Klebsiella pneumoniae complex TOC (Day 21): number analyzed (Participants) | 19 | 7
  Klebsiella pneumoniae complex TOC (Day 21) | 31.6 | 71.4
  Klebsiella pneumoniae complex LFU (Day 28): number analyzed (Participants) | 19 | 7
  Klebsiella pneumoniae complex LFU (Day 28) | 26.3 | 71.4
  Pseudomonas aeruginosa EOT (up to Day 14): number analyzed (Participants) | 13 | 3
  Pseudomonas aeruginosa EOT (up to Day 14) | 53.8 | 33.3
  Pseudomonas aeruginosa TOC (Day 21): number analyzed (Participants) | 13 | 3
  Pseudomonas aeruginosa TOC (Day 21) | 30.8 | 33.3
  Pseudomonas aeruginosa LFU (Day 28): number analyzed (Participants) | 13 | 3
  Pseudomonas aeruginosa LFU (Day 28) | 15.4 | 33.3
  Proteus mirabilis EOT (up to Day 14): number analyzed (Participants) | 1 | 2
  Proteus mirabilis EOT (up to Day 14) | 0.0 | 0.0
  Proteus mirabilis TOC (Day 21): number analyzed (Participants) | 1 | 2
  Proteus mirabilis TOC (Day 21) | 0.0 | 0.0
  Proteus mirabilis LFU (Day 28): number analyzed (Participants) | 1 | 2
  Proteus mirabilis LFU (Day 28) | 0.0 | 0.0
  Escherichia coli EOT (up to Day 14): number analyzed (Participants) | 1 | 1
  Escherichia coli EOT (up to Day 14) | 100.0 | 100.0
  Escherichia coli TOC (Day 21): number analyzed (Participants) | 1 | 1
  Escherichia coli TOC (Day 21) | 100.0 | 100.0
  Escherichia coli LFU (Day 28): number analyzed (Participants) | 1 | 1
  Escherichia coli LFU (Day 28) | 0.0 | 100.0
  Haemophilus influenzae EOT (up to Day 14): number analyzed (Participants) | 2 | 0
  Haemophilus influenzae EOT (up to Day 14) | 100.0 |
  Haemophilus influenzae TOC (Day 21): number analyzed (Participants) | 2 | 0
  Haemophilus influenzae TOC (Day 21) | 100.0 |
  Haemophilus influenzae LFU (Day 28): number analyzed (Participants) | 2 | 0
  Haemophilus influenzae LFU (Day 28) | 100.0 |
  Burkholderia cepacia complex EOT (up to Day 14): number analyzed (Participants) | 1 | 0
  Burkholderia cepacia complex EOT (up to Day 14) | 100.0 |
  Burkholderia cepacia complex TOC (Day 21): number analyzed (Participants) | 1 | 0
  Burkholderia cepacia complex TOC (Day 21) | 100.0 |
  Burkholderia cepacia complex LFU (Day 28): number analyzed (Participants) | 1 | 0
  Burkholderia cepacia complex LFU (Day 28) | 100.0 |
  Citrobacter freundii complex EOT (up to Day 14): number analyzed (Participants) | 1 | 0
  Citrobacter freundii complex EOT (up to Day 14) | 100.0 |
  Citrobacter freundii complex TOC (Day 21): number analyzed (Participants) | 1 | 0
  Citrobacter freundii complex TOC (Day 21) | 100.0 |
  Citrobacter freundii complex LFU (Day 28): number analyzed (Participants) | 1 | 0
  Citrobacter freundii complex LFU (Day 28) | 100.0 |
  Enterobacter cloacae complex EOT (up to Day 14): number analyzed (Participants) | 0 | 1
  Enterobacter cloacae complex EOT (up to Day 14) |  | 100.0
  Enterobacter cloacae complex TOC (Day 21): number analyzed (Participants) | 0 | 1
  Enterobacter cloacae complex TOC (Day 21) |  | 100.0
  Enterobacter cloacae complex LFU (Day 28): number analyzed (Participants) | 0 | 1
  Enterobacter cloacae complex LFU (Day 28) |  | 0.0
  Pseudomonas otitidis EOT (up to Day 14): number analyzed (Participants) | 1 | 0
  Pseudomonas otitidis EOT (up to Day 14) | 100.0 |
  Pseudomonas otitidis TOC (Day 21): number analyzed (Participants) | 1 | 0
  Pseudomonas otitidis TOC (Day 21) | 100.0 |
  Pseudomonas otitidis LFU (Day 28): number analyzed (Participants) | 1 | 0
  Pseudomonas otitidis LFU (Day 28) | 100.0 |
  Ralstonia pickettii EOT (up to Day 14): number analyzed (Participants) | 1 | 0
  Ralstonia pickettii EOT (up to Day 14) | 100.0 |
  Ralstonia pickettii TOC (Day 21): number analyzed (Participants) | 1 | 0
  Ralstonia pickettii TOC (Day 21) | 100.0 |
  Ralstonia pickettii LFU (Day 28): number analyzed (Participants) | 1 | 0
  Ralstonia pickettii LFU (Day 28) | 100.0 |
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; A.calco/baumannii complex EOT (up to Day 14); Test type: Other; Treatment difference = 30.3, 95% CI 2-sided [-4.2 to 64.8]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; A.calco/baumannii complex TOC (Day 21); Test type: Other; Treatment difference = 12.0, 95% CI 2-sided [-19.1 to 43.2]
Statistical Analysis 3: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; A.calco/baumannii complex LFU (Day 28); Test type: Other; Treatment difference = 0.5, 95% CI 2-sided [-29.0 to 29.9]
Statistical Analysis 4: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; EOT (up to Day 14); Test type: Other; Treatment difference = -8.3, 95% CI 2-sided [-57.9 to 41.1]
Statistical Analysis 5: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella pneumoniae complex TOC (Day 21); Test type: Other; Treatment difference = -39.8, 95% CI 2-sided [-89.1 to 9.4]
Statistical Analysis 6: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Klebsiella pneumoniae complex LFU (Day 28); Test type: Other; Treatment difference = -45.1, 95% CI 2-sided [-93.8 to 3.5]
Statistical Analysis 7: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Pseudomonas aeruginosa EOT (up to Day 14); Test type: Other; Treatment difference = 20.5, 95% CI 2-sided [-59.8 to 100.0]
Statistical Analysis 8: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Pseudomonas aeruginosa TOC (Day 21); Test type: Other; Treatment difference = -2.6, 95% CI 2-sided [-82.0 to 76.9]
Statistical Analysis 9: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Pseudomonas aeruginosa LFU (Day 28); Test type: Other; Treatment difference = -17.9, 95% CI 2-sided [-95.3 to 59.4]
Statistical Analysis 10: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; Escherichia coli LFU (Day 28); Test type: Other; Treatment difference = -100.0, 95% CI 2-sided [-100.0 to 0.0]

22. Secondary Outcome: The Percentage of Participants With Overall Success in the Micro-MITT Population
Description: Overall success was defined as clinical success and microbiological success at the visits of EOT or TOC, or sustained success for clinical outcome and microbiological success at the visit of LFU. Microbiological success included eradication or presumed eradication.
Time Frame: EOT (up to Day 14), TOC (Day 21), and LFU (Day 28)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 113 | 57
percentage of participants
  EOT (up to Day 14) | 75.2 | 64.9
  TOC (Day 21) | 50.4 | 47.4
  LFU (Day 28) | 47.8 | 40.4
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; EOT (up to Day 14); Test type: Other; Treatment difference = 10.2, 95% CI 2-sided [-4.9 to 25.3]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; TOC (Day 21); Test type: Other; Treatment difference = 3.0, 95% CI 2-sided [-13.0 to 19.0]
Statistical Analysis 3: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; LFU (Day 28); Test type: Other; Treatment difference = 7.9, 95% CI 2-sided [-7.6 to 23.5]

23. Secondary Outcome: The Percentage of Participants With Overall Success in the Extended Micro-MITT Population
Description: as for outcome 22
Time Frame: EOT (up to Day 14), TOC (Day 21), and LFU (Day 28)
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 153 | 78
Percentage of participants
  EOT (up to Day 14) | 68.6 | 61.5
  TOC (Day 21) | 45.8 | 44.9
  LFU (Day 28) | 42.5 | 39.7
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; EOT (up to Day 14); Test type: Other; Treatment difference = 7.5, 95% CI 2-sided [-5.8 to 20.8]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; TOC (Day 21); Test type: Other; Treatment difference = 1.9, 95% CI 2-sided [-11.6 to 15.5]
Statistical Analysis 3: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; LFU (Day 28); Test type: Other; Treatment difference = 4.1, 95% CI 2-sided [-9.2 to 17.4]

24. Secondary Outcome: The Percentage of Participants With Overall Success in the ME Population
Description: as for outcome 22
Time Frame: EOT (up to Day 14), TOC (Day 21), and LFU (Day 28)
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 96 | 51
Percentage of participants
  EOT (up to Day 14) | 78.1 | 72.5
  TOC (Day 21) | 57.3 | 52.9
  LFU (Day 28) | 54.2 | 45.1
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; EOT (up to Day 14); Test type: Other; Treatment difference = 4.8, 95% CI 2-sided [-10.6 to 20.2]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; TOC (Day 21); Test type: Other; Treatment difference = 3.2, 95% CI 2-sided [-14.0 to 20.4]
Statistical Analysis 3: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; LFU (Day 28); Test type: Other; Treatment difference = 8.6, 95% CI 2-sided [-8.4 to 25.6]

25. Secondary Outcome: The Percentage of Participants With Overall Success in the CR-MITT Population
Description: as for outcome 22
Time Frame: EOT (up to Day 14), TOC (Day 21), and LFU (Day 28)
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 53 | 23
Percentage of participants
  EOT (up to Day 14) | 47.2 | 34.8
  TOC (Day 21) | 22.6 | 26.1
  LFU (Day 28) | 17.0 | 26.1
Statistical Analysis 1: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; EOT (up to Day 14); Test type: Other; Treatment difference = 11.2, 95% CI 2-sided [-14.5 to 36.9]
Statistical Analysis 2: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; TOC (Day 21); Test type: Other; Treatment difference = -5.4, 95% CI 2-sided [-28.4 to 17.6]
Statistical Analysis 3: Comparison: Imipenem/Cilastatin and XNW4107 vs Imipenem/Cilastatin/Relebactam; LFU (Day 28); Test type: Other; Treatment difference = -10.2, 95% CI 2-sided [-32.9 to 12.5]

26. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A TEAE was defined as any untoward medical occurrence after first dose associated with the use of a drug in humans, whether or not considered drug-related. An SAE was defined as any adverse event (AE) occurring at any dose that met one or more of the following criteria: resulted in death, was life-threatening, required participant hospitalization or prolongation of an existing hospitalization, resulted in persistent or significant disability or incapacity, a congenital anomaly or birth defect or an important medical event.
Time Frame: Day 1 to Day 28
Population: Measured in the safety population, which included all participants who received at least 1 dose of study drug during the study. Participants were analyzed according to the treatment received during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
Number analyzed (Participants) | 299 | 150
Participants
  TEAE | 286 | 147
  SAE | 34 | 10

27. Secondary Outcome: Blood XNW4107, Imipenem, and Cilastatin Concentrations
Description: Blood samples were taken for analysis of XNW4107, imipenem, and cilastatin concentrations. The data at each time point was calculated as an average across Days 4, 5 and 6.
Time Frame: Predose, 5-25 minutes post-dose, and 2-3 hours post-dose on Day 4, 5, or 6
Population: Measured in the pharmacokinetic (PK) population, which included all participants from the safety population during the study with at least 1 reportable concentration of XNW4107, imipenem, or cilastatin. As pre-specified, data for PK was collected and reported only for the study drug treatment group (Imipenem/Cilastatin and XNW4107).
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/ml)
Arm/Group | Imipenem/Cilastatin and XNW4107
Number analyzed (Participants) | 286
nanograms per milliliter (ng/ml)
  XNW4107 Day (D)4/D5/D6 Pre-dose | 3840 (3330)
  XNW4107 D4/D5/D6 5-25min post dose | 16000 (6030)
  XNW4107 D4/D5/D6 2-3hour post dose | 7320 (3890)
  Imipenem D4/D5/D6 Pre-dose | 1770 (2050)
  Imipenem D4/D5/D6 5-25min post dose | 22900 (9310)
  Imipenem D4/D5/D6 2-3hour post dose | 5970 (2980)
  Cilastatin D4/D5/D6 Pre-dose | 1910 (3350)
  Cilastatin D4/D5/D6 5-25min post dose | 24200 (10100)
  Cilastatin D4/D5/D6 2-3hour post dose | 5610 (4720)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 28
Description: Measured in the safety population, which included all participants who received at least 1 dose of study drug during the study. Participants were analyzed according to the treatment received during the study.
Arm/Group | Imipenem/Cilastatin and XNW4107 | Imipenem/Cilastatin/Relebactam
All-Cause Mortality (participants affected / at risk) | 23/299 | 5/150
Serious Adverse Events (participants affected / at risk) | 34/299 | 10/150
Other Adverse Events (participants affected / at risk) | 260/299 | 136/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imipenem/Cilastatin and XNW4107 (N=299) | Imipenem/Cilastatin/Relebactam (N=150)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (2) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Gastric mucosal lesion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematological infection (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (2) | 0 (0)
Mydriasis (Eye disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 1 (3) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Brain stem syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Death (General disorders and administration site conditions) | 6 (6) | 0 (0)
Multiple organ dysfunction syndrome (General disorders and administration site conditions) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders and administration site conditions) | 1 (1) | 0 (0)
Brain herniation (Injury, poisoning and procedural complications) | 2 (2) | 2 (3)
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imipenem/Cilastatin and XNW4107 (N=299) | Imipenem/Cilastatin/Relebactam (N=150)
Hyponatraemia (Metabolism and nutrition disorders) | 97 (198) | 53 (101)
Hypokalaemia (Metabolism and nutrition disorders) | 109 (185) | 36 (61)
Hypoproteinaemia (Metabolism and nutrition disorders) | 76 (106) | 22 (37)
Hypocalcaemia (Metabolism and nutrition disorders) | 50 (94) | 13 (23)
Hypochloraemia (Metabolism and nutrition disorders) | 29 (48) | 14 (19)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 27 (44) | 13 (20)
Hypernatraemia (Metabolism and nutrition disorders) | 16 (26) | 10 (24)
Anaemia (Blood and lymphatic system disorders) | 123 (234) | 51 (98)
Constipation (Gastrointestinal disorders) | 50 (67) | 28 (52)
Diarrhoea (Gastrointestinal disorders) | 51 (60) | 26 (27)
Vomiting (Gastrointestinal disorders) | 22 (25) | 9 (10)
Alanine aminotransferase increased (Investigations) | 60 (110) | 40 (74)
Aspartate aminotransferase increased (Investigations) | 56 (106) | 37 (93)
Gamma-glutamyltransferase increased (Investigations) | 30 (46) | 14 (25)
Blood alkaline phosphatase increased (Investigations) | 15 (20) | 10 (15)
Venous thrombosis limb (Vascular disorders) | 30 (35) | 12 (17)
Deep vein thrombosis (Vascular disorders) | 23 (28) | 18 (20)
Urinary tract infection (Infections and infestations) | 50 (58) | 23 (29)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 22 (30) | 5 (9)
Rash (Skin and subcutaneous tissue disorders) | 16 (16) | 8 (9)
Hyperlipidaemia (Metabolism and nutrition disorders) | 17 (27) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT05204563/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT05204563/SAP_001.pdf